CLINICAL TRIAL: NCT06414421
Title: The Effect of Transcute Electrical Nerve Stimulation On Pain, Complication and Comfort in Patients Who Undergo Prostate Biopsy With Transrectal Ultrasound
Brief Title: The Effect of TENS on Pain, Complications and Comfort in Patients Who Had Prostate Biopsy With Transrectal Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Sevda Fırat, Principal Investigator, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CukurovaUSFırat
Record Dates: First submitted 2023-12-13; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer XXX
Keywords: Transcutaneous Electrical Nerve Stimulation (TENS)

STUDY DESIGN:
Intervention Model Description: This study was conducted as a two-group randomized controlled intervention study to determine the effect of TENS application on pain, complications and comfort in patients undergoing transrectal ultrasound-guided prostate biopsy (TRUSG-PBx).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS (Experimental): In TENS group patients, 4 electrodes of the TENS device (2 on the front side: on the anterior right and left groin skin, 2 on the back side: on the right and left presacral skin) were placed 3-5 minutes before the biopsy procedure, and the application was started and TENS was applied throughout the procedure. continued. TENS was applied again for 30 minutes 2 hours after the procedure. Frequency of the TENS program applied in the conventional model: 100 Hz; pulse width: 150 μs; duration:30 minutes; The current intensity (amplitude: highest level 60 mA) is adjusted (according to individual tolerance by asking the patient) to create a tingling or pricking sensation that does not disturb the patient.Data were collected in three stages.
  Interventions: Other: Transcuten Electriacal Nerve Stimulation
- CONTROL (No Intervention): TENS application was not performed. Data were collected in three stages. The first (before biopsy) and second (during and after biopsy) stages were carried out face to face, and the third stage (after discharge) was conducted by telephone interview technique.
  Research data; The data were collected by the researcher using face-to-face and telephone interview techniques using the "Personal Information Form", "Pain Evaluation Form", "TRUSG-PBx Complication Monitoring Form" and "Perianesthesia Comfort Scale", which evaluate the personal and disease-related characteristics of the patients.

INTERVENTIONS:
Other: Transcuten Electriacal Nerve Stimulation — In TENS group patients, 4 electrodes of the TENS device were placed 3-5 minutes before the biopsy procedure, and the application was started and TENS was applied throughout the procedure. continued. TENS was applied again for 30 minutes 2 hours after the procedure.
  Arms: TENS

SUMMARY:
Prostate cancer is one of the most common types of malignancy in men. Transrectal Ultrasound Guided Prostate Biopsy (TRUSG-PBx) is considered the gold standard method. The present, Transrectal ultrasound guided prostate biopsy is considered the gold standard method in the diagnosis of prostate cancer. During the process, patients experience severe discomfort and pain, although anesthetics and analgesics are used. In addition to pharmacological methods, non-pharmacological methods are also used in the control of pain caused by diagnosis and treatment interventions. Transcutaneous Electrical Nerve Stimulation (TENS) is among the non-pharmacological methods and it is the most widely used electroanalgesia method. In this randomized controlled intervention research, the effect of TENS application will be evaluated on pain, complications and comfort level during and after the procedure in patients who underwent Transrectal Ultrasound-Guided Prostate Biopsy. Thanks to this research, it is thought that the pain level and complications will decrease and the comfort level will increase in patients who undergo TENS application.

The research will be carried out in Çukurova University Faculty of Medicine Balcalı Application and Research Hospital Urology Outpatient Clinic. The sample of the research will create volunteer patients, providing research criteria and made prostate biopsy in Urology Outpatient Clinic. Patients consisting of 2 groups as control and experimental (TENS applied) will be determined by randomization. In the power analysis calculated with statistical support, confidence interval of 95%, alpha value 0.05, beta value calculated with 80% power, a total of 80 patients will be included in the control and experimental group, including 40 patients each. The data will be collected by "Personal Information Form", "Pain Assessment Form", "TRUSG-PBx Complication Follow-up Form", "Perianesthesia Comfort Scale Form". The data obtained will be analyzed in SPSS (Statisticial Package for the Social Sciences) package program.

In this context, our research, a comparison will be made by evaluating the effect of TENS application on pain, complications and comfort, in patients who underwent transrectal ultrasound-guided prostate biopsy. These results, non-pharmacological methods will make great contributions to improving patient outcomes in diagnostic interventions.

Keywords: Pain, Nurse, Comfort, Prostate Biopsy and Complications, Transcutaneous Electrical Nerve Stimulation (TENS).

DETAILED DESCRIPTION:
Prostate cancer is one of the most common types of malignancy in men. According to GLOBOCAN (Global cancer statistics) 2020 data, the age-standardized incidence rate of prostate cancer varies between 37.5-11.3 per hundred thousand in the world, depending on the development level of the countries, and it is seen to be 42.5 per hundred thousand in our country. It ranks second after lung cancer in terms of incidence in men in our country and in the world.

Prostate cancer screening aims to reduce mortality and morbidity by detecting prostate cancer at an early stage. In the diagnosis of prostate cancer, digital rectal examination (DRE), prostate specific antigen (PSA) value, transrectal ultrasonography (TRUSG) and biopsy are used.

Transrectal ultrasound-guided prostate biopsy (TRUSG-PBx) is currently considered the gold standard method in the diagnosis of prostate cancer.

In the TRUSG-guided biopsy procedure, patients are placed in the left lateral or lithotomy position, a needle-guided rectal probe is inserted into the anal canal with the help of lubricating gel, and the prostate tissue is monitored under ultrasound guidance and a biopsy is taken. The procedure takes approximately 20-30 minutes, and insertion and removal of the probe into the rectal area takes approximately 10-15 minutes in total.

TRUSG-PBx is a cost-effective, accessible invasive procedure that has undergone significant changes and developments over the years, is well tolerated, has minimally serious, undesirable side effects and complications, can be easily and quickly performed in outpatient conditions. However, although it is a safe method with a low complication rate, each patient must be carefully monitored because it is an invasive procedure. Complications frequently include hematuria, hematospermia, rectal bleeding, dysuria, urinary retention, hematochezia, erectile dysfunction, infection, prostatitis and pain. In most patients who will undergo transrectal biopsy, the possibility of the result being cancer and the psychological discomfort caused by the fact that the procedure will be performed rectally increase the pain.

Although prostate biopsy is thought to be well tolerated by patients, it appears to cause discomfort and pain in 65% to 90% of cases. Failure to recognize and deal with this problem not only affects patients' willingness to undergo the procedure again if necessary, but can also potentially lead to forgoing prostate evaluation or rejection of the procedure for fear of a painful invasive procedure. In addition, the importance of pain control has gradually increased due to prostate biopsy being performed on younger patients, biopsies being taken from more quadrants, and repeated prostate biopsies. Due to severe pain, the rate of tolerance of the procedure by the patient decreases, and this may lead to a decrease in the number of biopsy samples taken from the planned quadrant and a decrease in cancer detection rates. Therefore, it is extremely important to ensure pain control and increase patient tolerance and comfort in TRUSG-PBx.

The pain felt during the biopsy occurs for 2 reasons. The first is pain caused by stretching of the anal sphincter as the transrectal ultrasound probe enters the anus (passing the ultrasound probe through the anus, advancing it into the rectum, and manipulating it within the rectum). Especially before biopsy, periprostatic nerve blockade requires penetration into the rectum with a rectal probe before anesthesia, and this first penetration causes the patients' complaints. The second is the pain felt when the biopsy needle penetrates the prostate capsule and enters the prostatic stroma.

Pharmacological methods such as local anesthetics, peripheral nerve blockade, spinal and intravenous (IV) sedation applications have been used to reduce pain and discomfort, and results have been reported showing that these methods increase pain tolerance in the patient. The increasing use of active surveillance and the acceptance of prostate biopsy for prostate cancer management are very important to relieve or reduce patients' discomfort during biopsy and optimize satisfaction and comfort.

Although TRUSG-PBx is easy to perform and causes very low mortality, there is a need to develop new protocols for analgesia before the procedure to reduce the discomfort and pain that patients may feel.

Nurses should also apply non-pharmacological methods to reduce the consumption of analgesic drugs or increase their effect by providing adequate analgesia. Nurses, who have a key role in the pain management team, should do what is necessary about pain preventive approaches and pain control methods at this stage.

Non-pharmacological methods are important in providing comfort and a feeling of control, improving functionality and quality of life, and reducing pain and anxiety.

TRUSG-PBx is a challenging diagnostic procedural intervention due to pain and fear for patients. For this reason, non-pharmacological methods should be used and pharmacological methods should be integrated into nursing practices in order to tolerate the procedure by patients and ensure effective pain control.

Among the non-pharmacological methods that can be used safely in acute painful interventions, Transcutaneous Electrical Nerve Stimulation (TENS) is an effective electroanalgesia method. This method is a method of applying controlled low-voltage electrical current to the nervous system through electrodes placed on the skin. The pain-relieving effect of TENS is explained in two ways. The first is that TENS stimulates the sensory A fibers with high frequency stimulation, and the impulses of this stimulation cover the path to the brain and close the door to the passage of pain. Secondly, it affects the perception of pain by initiating the release of natural opioids in the body. It is widely used in acute and chronic pain. TENS is an analgesia method requested by the specialist doctor. How TENS will be applied to which patient, its parameters, application area and duration are determined by the doctor, and it requires the cooperation of a nurse trained in TENS (from a physiotherapy or algology specialist in TENS application) and the doctor. Many studies in this field show that TENS reduces pain.

Although there are many evidence-based studies in the literature on pharmacological methods that reduce pain in TRUSG-PBx, the number of studies on non-pharmacological methods is quite limited.

Our clinical examinations show that non-pharmacological methods are used very rarely in TRUSG-PBx, there is no protocol to reduce pain during and after biopsy, and nurses do not apply TENS. Additionally, no studies have been found in the literature regarding the effect of TENS application on pain, complications and comfort during and after TRUSG-PBx. This study will guide nurses in using and developing non-pharmacological methods in clinics, choosing the appropriate ones for patients with their positive and negative aspects, evaluating their effectiveness, contributing to the professional and independent roles of the nursing profession, increasing the quality of care and providing comfort and satisfaction, thereby increasing the feeling of professional satisfaction. It is thought that it will increase. In addition, it will contribute to the effective application of TENS, which is a simple, cheap and effective method that nurses, who are responsible for patient follow-up and treatment, provide direction and provide uninterrupted health services, have the authority to apply together with the physician, and will guide the development of non-pharmacological analgesia applications. It is thought that nonpharmacological methods will improve patient outcomes in the control of procedural pain resulting from diagnostic interventions.

Purpose of the research:

This study was conducted to determine the effect of TENS on pain, comfort level and complications in patients who underwent transrectal ultrasound-guided prostate biopsy.

ELIGIBILITY:
Inclusion Criteria:

* • Able to communicate,

  * Those who are over 40 years old,
  * Being literate,
  * No previous history of chronic pain,
  * Not addicted to alcohol or drugs,
  * Without bleeding diathesis and active urinary tract infection,
  * Having no cognitive impairment, neurological or psychiatric disease,
  * Do not have any inflammatory rheumatological, neurological or cognitive disease,
  * No contraindications for electrotherapy (pacemaker, arrhythmia, epilepsy, dermatological diseases),
  * Not using chronic opioids, antidepressants or psychoactive drugs,
  * Those who have not had TENS application before,
  * No skin lesions in the electrode connection areas,
  * No significant anorectal disease (wound, fistula, fissure, hemorrhoids, etc.),
  * As a result of the evaluation by the physician, there is no harm in applying TENS,
  * Patients who voluntarily agreed to participate in the research were included.

Exclusion Criteria:

* Lidocaine gel was applied to the anal area and rectum before the biopsy, or a different anesthetic method was used (IV, IM, rectal anesthetic/analgesic drug application or general anesthesia, etc.),
* Coming for prostate biopsy followed by Foley catheter,
* Patients who did not agree to participate in the research were not included in the sample.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — prostate
Enrollment: 80 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Pain Scale (Numerical pain scale) | The first 24 hours: NPS 1, 2, 3, 4, 5, 6, 7, 8, 9
  The scale used in the first part of this form, which is intended to evaluate pain severity, is the Numerical Pain Scale (NPS). On this scale, it starts with absence of pain (0) and reaches the level of unbearable pain (10).According to the determined measurement times of the patients [T1: At the beginning of the biopsy/while the ultrasound probe is being placed (NPS-1), T2: During the biopsy/5 minutes after the ultrasound probe is placed (NPS-2), T3: At the end of the biopsy/while the ultrasound probe is being removed (NPS-3). , T4: 1 hour after the end of the biopsy (NPS-4), T5: 2 hours after the end of the biopsy (NPS-5), T6: 2.5 hours after the end of the biopsy (NPS-6), T7: During the first urination after the biopsy (NPS-6). -7), T8: 6 hours after the end of the biopsy (NPS-8), T9: 24 hours after the end of the biopsy (NPS-9)]. The second part of the pain evaluation form includes information about the analgesic medication used in the first 6 and 24 hours.

SECONDARY OUTCOMES:
Complication (TRUSG-PBx Complication Monitoring Form) | Hematuria, hematospermia, rectal bleeding, urinary retention, dysuria, anal pain seen in the first 24 hours and 1 week
  Comparison of complications of patients according to time Prepared by the researchers in line with the literature, the first part of TKIF, prepared by the researchers in line with the literature, aims to determine bleeding during biopsy (rectal bleeding, bleeding from the urethra) and bleeding in the first urine after biopsy, and the second part / after discharge (at home) aims to determine complications that may develop after biopsy. 6 items are included (hematuria, hematospermia, rectal bleeding, dysuria, anal pain, urinary retention).

OTHER OUTCOMES:
Comfort (Perianesthesia Comfort Scale (PCS) | Comparison of patients' Perianesthesia Comfort Scale (PCS) scores in the first 24 hours
  The scale consists of 24 items and questions the individual's feelings, thoughts and feelings before and after the surgical procedure. Each item in the scale is a Likert type with a score ranging from 1 to 6 points, from "strongly disagree" to "strongly agree". It consists of positive and negative substances. 12 of the items are positive and 12 are negative.Negative statements are reversed when scoring.Accordingly, in positive items, a high score (6) indicates high comfort, a low score (1) indicates low comfort, and in negative items, a low score (1) indicates high comfort and a high score (6) indicates low comfort. In the evaluation of the scale; The resulting negative scores are reverse coded and summed with positive scores. The highest score that can be obtained from the scale is 144 and the lowest score is 24. As a result, as the score increases, comfort increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Sariçam, Turkey (Türkiye)